CLINICAL TRIAL: NCT06833346
Title: BASICS: Back-pain Alleviation Via a Specific and Inexpensive Contextual Strength Training Protocol
Brief Title: Efficacy of Hip Belt Squat Training on Pain Management and Physcial Function in Low Back Pain Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Aleris (Unknown)
Responsible Party: Principal Investigator, Mathias Kristiansen, Associate Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20230063-B
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Low back pain patients not performing an intervention
- Hip belt squat exercise (Experimental): Low back pain patients performing hip belt squat training twice per week for 12 weeks.
  Interventions: Other: Hip belt squat exercise

INTERVENTIONS:
Other: Hip belt squat exercise — Hip belt squat exercise performed twice per week for 12 weeks
  Arms: Hip belt squat exercise

SUMMARY:
The purpose of this project is to investigate the efficacy of the hip belt squat exercise in pain management and physical function for people with chronic low back pain.

DETAILED DESCRIPTION:
This study is a randomized controlled trial (RCT) designed to evaluate the effectiveness of a 12-week hip belt squat (HBS) intervention for patients with non-specific low back pain (LBP). Participants, aged 18-60 with LBP for more than 12 weeks, are randomly assigned to either the intervention group or a control group. The control group will not receive any intervention, whereas the HBS intervention consists of two supervised sessions per week for 12 weeks, with load adjustments based on perceived exertion.

The study aims to recruit 50-60 patients to ensure sufficient statistical power. Primary outcomes include health-related quality of life (EQ-5D-5L), fear-avoidance beliefs (FABQ), functional ability (ODI), risk of chronicity (STarTBack), pain intensity (VAS), and pain sensitivity (PPT). Secondary outcomes include body composition (DEXA), lumbar flexibility, maximal muscle strength (5RM), physical activity (GPAQ), tobacco use (SQ), and work-related stress (WSQ).

Measurements are taken at baseline, 6 weeks, 12 weeks, and a 1-year follow-up for various outcomes. This comprehensive approach aims to provide valuable insights into the effectiveness of the HBS intervention for managing LBP.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with non-specific low back pain for more than twelve weeks, with a VAS score of at least 3, taken as an average of the last week, and ODI>20

Exclusion Criteria:

* Leg pain greater than back pain
* Neuromuscular disorders
* Spinal or lower extremity fractures
* Infections
* Cancer
* Osteoporosis
* Dementia
* Current substance abuse
* Former lumbar surgery
* Persistent pain syndromes other than back pain
* Inflammatory rheumatic diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Oswetry Disability index | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  A questionnaire measuring the degree of disability, which ranges from 0 (no disability) to 100 (bedridden).
Health related quality of life | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  A questionnaire measuring the easured health-related quality of life (EuroQOL-5D), ranging from -0.596 to 1, with higher scores indicating better quality of life.
Fear-avoidance Beliefs Questionnaire | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  Fear-avoidance Beliefs Questionnaire (FABQ) measuring the amount of kinesiophobia, ranging from 0-96 with higher scores indicating higher levels of fear avoidance belief.
STarTBack tool | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  A questionnaire used to assess the risk of chronicity in low back pain (ranging from low to medium to high risk).
Pain sensitivity | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  Pressure-pain threshold was assessed using a handheld pressure algometer.
Pain intensity | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  Patients were asked to rate the intensity of their LBP on a visual analog scale (VAS) using a 10 cm long line, where the far-left part of the line (0/10) corresponded to no pain and the far right part (10/10) corresponded to the worst imaginable pain. Ratings on the VAS scale was gathered both while the participants stood in an upright position and during a self-chosen movement known to induce pain (e.g. bending over).

SECONDARY OUTCOMES:
Muscle strength | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  Muscle strength was assessed in the hop belt squat exercise using a 5 repetition maximum test
Lumbar flexibility | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  Lumbar flexibility was assessed using a custom made test.
Body composition | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  To assess changes in body composition a DEXA scan was performed. This test quantified lean body mass (kg) and fat mass (kg).
Physical activity level | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  To assess the physical activity level of the patients the Global Physical Activity Questionnaire (GPAQ) questionnaire was used.
  Higher scores indicate higher levels of physical activity, which is considered better for health. Lower scores indicate lower levels of physical activity, which is considered worse for health.
  Interpretation: High Physical Activity: More than 3000 MET-minutes per week. Moderate Physical Activity: Between 600 and 3000 MET-minutes per week. Low Physical Activity: Less than 600 MET-minutes per week.
Tobacco use | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  To assess tobacco use, patients were questioned using the Smoking Questionnaire (SQ).
Work related stress | Assessed at baseline, after 6 weeks, 12 weeks, and at 1-year followup
  To assess work related stress, the Work Stress Questionnaire (WSQ) was used.
  Lower scores indicate lower levels of work-related stress, which is considered better for overall well-being.
  Higher scores indicate higher levels of work-related stress, which can negatively impact health and job performance.
  Interpretation:
  Scores below 135: Indicate a normal level of work-related stress. Scores of 135 or above: Suggest an unusual amount of work-related stress, indicating the need for stress management interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data is protected under GDPR